CLINICAL TRIAL: NCT00020098
Title: Use of Complementary or Alternative Medicine Practices by Women at Increased Risk for Breast Cancer
Brief Title: Complementary or Alternative Medicine Practices Used by Women at Increased Risk for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Prevention
Other Study IDs: 000039; 00-C-0039; MB-NAVY-B99-088; CDR0000067716
Record Dates: First submitted 2001-07-11; First posted 2004-02-27 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Procedure: evaluation of cancer risk factors

SUMMARY:
RATIONALE: Increasing knowledge about the complementary or alternative medicine practices used by women who are at increased risk for breast cancer may provide useful information for planning breast-cancer-prevention strategies.

PURPOSE: Clinical trial to determine how many women who are at increased risk for breast cancer use complementary or alternative medicine.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the prevalence of complementary or alternative medicine (CAM) practices among adult women who are enrolled in the Risk Assessment Clinic at the National Naval Medical Center Breast Care Center and are found to be at increased risk for developing breast cancer. II. Correlate the use of CAM with individual risk for breast cancer. III. Define the types of CAM practices used by this study population. IV. Identify reasons why this study population is using CAM.

OUTLINE: Patients are stratified according to prevalence of complementary and alternative medicine practices (enteral/parenteral vs psychologic/neurologic). Patients complete a Personal Risk Assessment form, pre-test/post-test knowledge questionnaires, and a survey questionnaire.

PROJECTED ACCRUAL: A total of 102 patients will be accrued for this study within approximately 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Enrolled in the Risk Assessment Clinic (RAC) of the National Naval Medical Center and found to be at increased risk for breast cancer based on at least one of the following: Estimated risk of at least 1.7% for developing breast cancer over the next 5 years, as determined by the Breast Cancer Risk Assessment Tool (BCRAT) Prior history of lobular carcinoma in situ or ductal carcinoma in situ Family history of breast or ovarian cancer consistent with autosomal dominant pattern of inheritance or empirically elevated risk of breast cancer based on a single first- or second-degree relative with breast or ovarian cancer Must have attended the RAC education session within past 3-6 months Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: Not specified Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No other prior cancer except ductal carcinoma in situ or basal cell carcinoma Able to read and understand English

PRIOR CONCURRENT THERAPY: Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Study Completion 2001-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Glauber, RN, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Naval Medical Center, Bethesda, Maryland
  - Medicine Branch, Bethesda, Maryland